CLINICAL TRIAL: NCT05731635
Title: Plantar Pressure Values in Patients With Ankylosing Spondylitis and Their Relation With Clinical and Radiological Parameters
Brief Title: Plantar Pressure Values in Patients With Ankylosing Spondylitis
Status: Completed | Type: Observational
Sponsor: Amasya University (Other)
Responsible Party: Principal Investigator, Esra Topçu, specialist doctor (esra topcu), Amasya University
Other Study IDs: 159
Record Dates: First submitted 2023-01-26; First posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Device is Used for Evalution (Event)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: plantar pressure values — Walking enables for extremely accurate and pointwise ground response force measurement because to plantar pressure measurement (pedobarography). It allows for the objective comparison and evaluation of the dynamic pressure put on the ground by the foot in contact with it. It is often used in clinics to assess foot mechanics and associated disorders that affect the foot sole. Additionally, plantar pressure analysis is useful for identifying, treating, and monitoring conditions that impact the lower extremity's axial alignment.

SUMMARY:
this study was discovered that clinical and radiological characteristics were related to plantar pressure assessments in patients with AS.

DETAILED DESCRIPTION:
Determine the correlation between the plantar pressure readings of AS patients and the clinical and radiological measures utilized in the monitoring of the condition.

Method: This study covered 75 participants. The quality of life was measured using ASQoL, BASMI, BASFI, and BASDAI, and demographic information was also recorded. The pedobarographic evaluations included the recording of static and dynamic plantar pressures

ELIGIBILITY:
Inclusion Criteria: patients diagnosed with AS -

Exclusion Criteria: Patients with cognitive dysfunction, vision loss that would prevent walking on the pedobarography platform, history of surgery and neurological deficit in the lower extremity, and patients who could not walk independently

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Seventy-five adult patients who applied to Celal Bayar University outpatient clinics and were diagnosed with AS according to the modified New York criteria were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2011-12-01 (Actual); Primary Completion 2012-12-01 (Actual); Study Completion 2012-12-01 (Actual)

PRIMARY OUTCOMES:
Pedobarographic Measurements | at begining
  The cases' foot sole pressures were measured using a pedobarography device of the RsScan International brand (1m, 3D Scientific+Balance software model). This technology measures both static (when standing) and dynamic foot sole pressures (walking). The device's pressure measuring platform has an overall frame size of 1068x418x12 mm, 8192 sensors totaling 4 sensors per cm2, and a sensor area of 975x325 mm. It has a 500 Hz frequency, a 0-200 N/cm2 pressure range, a 15° to 40° C temperature range, and a 220/110 volt connecting power.

IPD SHARING:
Plan to Share IPD: Undecided